CLINICAL TRIAL: NCT01189591
Title: Slow-wave Sleep Deprivation as a Possible Treatment for Major Depressive Disorder
Brief Title: Slow-wave Sleep Deprivation in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2013-0019; P20MH077967 NIH grant number; H-2007-0150 (Other: UW IRB); P20MH077967 (NIH)
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep deprivation (Experimental): Slow-wave sleep deprivation for one night as an experimental treatment for major depressive disorder
  Interventions: Device: Slow-wave deprivation

INTERVENTIONS:
Device: Slow-wave deprivation — Using acoustic tones to suppress slow-wave sleep

SUMMARY:
Sleep deprivation can acutely reverse depressive symptoms in patients with major depression. Although underlying mechanisms of the antidepressant action in sleep deprivation are unclear, many of these observations can be explained by abnormal slow wave homeostasis. This study will test the prediction that selectively reducing slow waves during sleep (slow wave deprivation; SWD), without disrupting total sleep time, will yield an antidepressant effect.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Among the inclusion criteria will be:

  * age range 18-35 years
  * right handedness
  * major depressive disorder according to DSM-IV (Diagnostic and Statical Manual-Revision 4) criteria (as determined by the Structured Clinical Interview for Diagnostic and Statical Manual-Revision 4), with Hamilton Rating Scale for *Depression scores of at least 18 on the first 17 items
  * no psychotropic medications for at least 4 weeks
  * no joint and muscular di
  * normal hearing
  * regular bedtimes and sleep duration, no time zone shifts in the last three weeks.

Exclusion Criteria:

* Diabetes requiring insulin treatment
* A serious heart disorder or subjects who have had a heart attack within the last 3 months
* A diagnosis of cancer in the past 3 years and/or has active neoplastic disease
* Clinically significant abnormalities on pre-study physical exam or physician evaluation
* Subjects who meet DSM-IV (Diagnostic and Statical Manual-Revision 4) criteria for alcohol/drug abuse problems within the last six months or are currently using illegal drugs.
* Female subjects of child-bearing potential who are pregnant or planning to become pregnant.
* Women of child-bearing must be practicing a medically acceptable form of birth control.
* Women of childbearing potential will be questioned about pregnancy status and form of birth control to be used at each visit.
* Women who are unsure of their pregnancy status will be given a urine pregnancy test.
* Subjects taking investigational medications
* Subjects currently undergoing electroconvulsive therapy (ECT) or therapeutic transcranial magnetic stimulation (TMS).
* Subjects who regularly perform night or late evening shift work (e.g. - "second" or "third" shifts) or have had travel with time zone shifts >3h in the last 3 weeks

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale | 24 hours

SECONDARY OUTCOMES:
Inventory of Depressive Symptomology | 24 hours
  rating scale of mood

CONTACTS AND LOCATIONS:
Overall Officials: Ruth M Benca, M.D., Ph.D, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Wisconsin Center for Sleep Medicine and Research, Madison, Wisconsin, United States